CLINICAL TRIAL: NCT04839796
Title: A Cohort Study on Disease Prevention and Health Promotion in Northeastern Region of Taiwan
Brief Title: Northeastern Taiwan Community Medicine Research Cohort
Acronym: NTCMRC
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201800289A3
Record Dates: First submitted 2021-03-28; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-01

CONDITIONS: Cohort Study
Keywords: NTCMRC; Maintenance Project; Health Care Activities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Participants residing in urban areas: Urban residents enjoy convenient transportation, have access to abundant medical resources, have more job opportunities, and are on average younger but are also exposed to more air pollution.
- Participants residing in rural areas: Rural residents have less access to transportation, medical resources, and job prospects comparatively and are comparatively older. However, Rural residents are exposed to less pollution in general.

SUMMARY:
The cohort study on disease prevention and health promotion in the northeastern region of Taiwan is a trial dedicated to large-scale generational research in northeastern Taiwan beginning in the August of 2013. The program aims to develop a comprehensive and integrated approach to disease prevention and community health. The researcher's cohort organizes healthcare outreaches for participants over the age of 20 residing in 64 administrative areas in Keelung city and new Taipei city. The researcher's sessions include a comprehensive health examination, health-related questionnaires, and disease awareness seminars.

Biological samples, questionnaire information, and medical data obtained from researcher's participants are stored in researcher's core laboratory. Depersonalized data and samples are shared with partnering trials approved by the Chang Gung Memorial Hospital Institutional review board. The investigators are currently partnered with 18 clinical trials spanning across multiple disciplines such as urology, hepatology, metabolism, physical therapy, and psychology.

DETAILED DESCRIPTION:
The cohort study on disease prevention and health promotion in the northeastern region of Taiwan is a trial dedicated to large-scale generational research in northeastern Taiwan beginning in the August of 2013. The program aims to develop a comprehensive and integrated approach to disease prevention and community health. The researcher's cohort organizes healthcare outreaches for participants over the age in Keelung city and new Taipei city. The researcher's sessions include a comprehensive health examination, health-related questionnaires and disease awareness seminars.

Biological samples, questionnaire information, and medical data obtained from the researcher's participants are stored in the researcher's core laboratory. Depersonalized data and samples are shared with partnering trials approved by the Chang Gung Memorial Hospital Institutional review board. The investigators are currently partnered with 18 clinical trials spanning across multiple disciplines such as urology, hepatology, metabolism, physical therapy, and psychology.

The investigators are also a member of the national "Establish Multi-omics Database of Smart Healthcare for Obesity Therapeutics involving " joint project and the national "Remote Medical Monitoring System-Linking Healthcare Industrial Ecosystem-Taiwanese Novel Disease Monitoring Solution" initiative.

Introduction: This research is conducted in the form of community health care activities. Through regular community health household activities, community residents' awareness of health is improved, and various pathogenic factors are analyzed to strengthen health education, improve living habits, reduce risk factors, and promote the health of community residents.

Project purpose: In order to promote community fitness, The investigators will conduct long-term community medicine generation research. This research consists of a series of collaborative projects such as chronic kidney disease, chronic liver disease, metabolic syndrome, depression, dementia, obesity, exercise rehabilitation, etc.

In community health care activities, collect biological samples such as blood, urine, feces, etc., as well as questionnaire data. This project will link participants relevant health data to establish a database for the generation of Keelung Chang Gung community medicine research. These data will be provided for analysis of co-operative plans related to generations of research and long-term tracking of participants health.

ELIGIBILITY:
Inclusion Criteria:

1. Residing in Keelung city and new Taipei city.
2. Mobile health and mental health
3. Participating in healthcare outreaches

Exclusion Criteria:

1. Under 20 years old
2. Participant without judgment
3. Participant has HIV

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who enroll in these community health activities and meet the following conditions:
  1. Over the age of 20.
  2. Residing in 64 administrative areas in Keelung city and new Taipei city.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2043-08 (Estimated); Study Completion 2043-08 (Estimated)

PRIMARY OUTCOMES:
Participant died during the observation period. | From 2013 Augus to Feb 2021
  Investigators keep in touch with participants and invite them to participate in healthcare outreaches every year.
Dementia | From 2013 Augus to Feb 2021
  The AD8 dementia screening interview is used to detect the early signs of dementia. Using the items in the form to check whether participants have similar symptoms, so as to detect and treat them as soon as possible.
Chronic Kidney Disease | From 2013 Augus to Feb 2021
  Chronic kidney disease is a type of kidney disease in which there is gradual loss of kidney function over a period of months to years.
Liver cancer | From 2013 Augus to Feb 2021
  Participant suffers from liver cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chiau Shyu, PHD, Principal Investigator — Community Medicine Research Center,Chang Gung Memorial Hospital,Keelung branch
Locations (1):
- Community Medicine Research Center Chang Gung Memorial Hospital Keelung,Taiwan,204, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu PW, Yeh CH, Lo CJ, Tsai TH, Chan YH, Chou YJ, Yang NI, Cheng ML, Sheu WH, Lai CC, Sytwu HK, Tsai TF. Trans-omics analyses identify the biochemical network of LPCAT1 associated with coronary artery disease. Biomark Res. 2025 Aug 20;13(1):107. doi: 10.1186/s40364-025-00821-y. PMID 40830908
- [Derived] Wei YC, Chen CK, Lin C, Shyu YC, Chen PY. Life After Traumatic Brain Injury: Effects on the Lifestyle and Quality of Life of Community-Dwelling Patients. Neurotrauma Rep. 2024 Mar 1;5(1):159-171. doi: 10.1089/neur.2023.0113. eCollection 2024. PMID 38463415
- [Derived] Wu IW, Tsai TH, Lo CJ, Chou YJ, Yeh CH, Cheng ML, Lai CC, Sytwu HK, Tsai TF. Discovery of a Biomarker Signature That Reveals a Molecular Mechanism Underlying Diabetic Kidney Disease via Organ Cross Talk. Diabetes Care. 2022 Jun 2;45(6):e102-e104. doi: 10.2337/dc22-0145. No abstract available. PMID 35546525